CLINICAL TRIAL: NCT03183388
Title: Brain Emotion Circuitry-Targeted Self-Monitoring and Regulation Therapy (BE-SMART)
Acronym: BE-SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0407026910; R61MH111929 (NIH); 3UG3MH111929-02S1 (NIH)
Record Dates: First submitted 2017-06-08; First posted 2017-06-12 (Actual); Results first posted 2024-02-29 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Mood Disorders
Keywords: psychotherapy
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Intervention Model Description: It is planned that 72 of the 86 participants who meet criteria for bipolar disorder (BDI, BDII, BD-OS) will complete this combined psychotherapy (BE-SMART) and imaging study. There will be variation of therapies, but no comparison between groups. Actigraphy and ecological momentary assessments on 20 participants will be integrated as part of the supplement to parent grant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BE-SMART (Experimental): Psychobehavioral intervention with focus either on teaching emotional regulation skills or regularizing daily sleep and activity levels.
  Interventions: Behavioral: BE-SMART

INTERVENTIONS:
Behavioral: BE-SMART — Participants will take part in 12 therapy sessions, at a rate of about 1 session every one to two weeks. Sessions are anticipated to last about 1 hour each. Sessions may be focused on teaching skills to regulate emotions or regularize sleep and activity. These therapy sessions may be videotaped and audiotaped (only with the expressed written consent of the participant, and when appropriate, the participant's parent or guardian). Participants will be asked to complete worksheets and practice the skills learned from these sessions and will be asked questions about feelings. There will be an interview, assessments and scanning performed prior to treatment and at the midpoint and end to assess progress. The intervening 9 sessions may be by video telecommunication. Participants may be given devices to track actigraphy and ecological momentary assessments.

SUMMARY:
New treatments to help to reduce the emotional dysregulation of mood disorders are critically needed. This is a study of an emotional dysregulation psychotherapy treatment in which participants will learn skills to help to down-regulate maladaptive emotional responses and learn beneficial, healthy habits. Investigators will perform symptom and behavioral assessments and scanning prior to the treatment and will then repeat scanning, symptom and behavioral assessments at the midpoint, and after the psychotherapy is completed. This collected information will assess whether the treatment can improve functioning of emotion regulation brain circuitry.

DETAILED DESCRIPTION:
Aim: To use functional magnetic resonance imaging (fMRI), before, at mid point, and after an emotional regulation intervention, to assess intervention-associated changes in brain circuitry responses to emotional stimuli.

Hypothesis : The emotional regulation psychotherapy treatment will be associated with changes in emotional regulation circuitry.

At the time of registration, the primary outcome "Changes in Functioning of Emotional Brain Circuitry" was the only outcome registered. This outcome is comprised of multiple measurements and was split up individually at the time of results entry and the original primary outcome measure was deleted.

ELIGIBILITY:
Inclusion Criteria:

* participants meeting Diagnostic and Statistical Manual Fifth Edition (DSM-5) criteria for BDI, BDII or BD Other Specified Bipolar (BD-OS).
* participants with mood symptoms, such as Hamilton Depression Rating Scale (Ham-D) score ≥ 15 and/or for hypomania/mild mania such as Young Mania Rating Scale (YMRS) ≥ 12.

Exclusion Criteria:

* history of significant medical illness, particularly illness associated with possible changes in cerebral tissue or cerebrovasculature (e.g. hypertension)
* history of neurologic abnormality, including significant head trauma (defined by loss of consciousness of ≥5-minutes duration), seizure disorder, cerebrovascular or neoplastic lesion, or neurodegenerative disorder.
* contraindication to MRI scanning, e.g. presence of a ferromagnetic object, including orthodontic braces, or claustrophobia.
* intelligence quotient (IQ) lower than 70
* pregnancy
* alcohol/substance use may be permitted if participant does not meet for DSM-5 current use disorder but will not be permitted for illicit substance use in the week prior to study.

Ages: 16 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hilary P Blumberg, MD, Principal Investigator — Yale University
Locations (1):
- Mood Disorders Research Program, Yale School of Medicine, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kim JA, Sankar A, Marks R, Carrubba E, Lecza B, Quatrano S, Spencer L, Constable RT, Pittman B, Lebowitz ER, Silverman WK, Swartz HA, Blumberg HP. Chronotherapeutic intervention targeting emotion regulation brain circuitry, symptoms, and suicide risk in adolescents and young adults with bipolar disorder: a pilot randomised trial. BMJ Ment Health. 2025 Feb 19;28(1):e301338. doi: 10.1136/bmjment-2024-301338. PMID 39971594

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 76 participants were enrolled and 60 started
Groups:
- BE-SMART DR: Adolescents and young adults with BD who received baseline scan and Brain Emotion Circuitry Targeted Self-Monitoring Regulation Daily Rhythms (BE-SMART DR)
- BE-SMART ER: Adolescents and young adults with bipolar disorder (BD) who received baseline scan and Brain Emotion Circuitry Targeted Self- Monitoring Regulation Therapy Emotion Regulation (BE-SMART ER)
Period: Overall Study
Arm/Group | BE-SMART DR | BE-SMART ER
Started | 30 | 30
Completed Mid-point | 20 | 19
Completed Participation in Intervention and Endpoint Assessment | 19 | 16
Completed All Procedures Including Endpoint Imaging | 17 | 14
Completed | 17 | 14
Not Completed | 13 | 16
Not completed — Lost to Follow-up | 3 | 5
Not completed — Physician Decision | 1 | 4
Not completed — Withdrawal by Subject | 4 | 1
Not completed — Moved | 1 | 0
Not completed — Met Exclusion Criteria | 2 | 2
Not completed — COVID Pandemic Related | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- BE-SMART ER: Adolescents and young adults with BD who received baseline scan and Brain Emotion Circuitry Targeted Self- Monitoring Regulation Therapy Emotion Regulation (BE-SMART ER)
- Total: Total of all reporting groups
Arm/Group | BE-SMART ER | BE-SMART DR | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 7 | 11
  Between 18 and 65 years | 26 | 23 | 49
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 20 | 39
  Male | 11 | 10 | 21
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 9
  Not Hispanic or Latino | 27 | 24 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 3 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 23 | 21 | 44
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Functional Magnetic Resonance Imaging (fMRI) Blood Oxygen-level Dependent (BOLD) Signal Changes in Left Amygdala at Baseline and at the End of the Intervention
Description: FMRI was performed during an emotional face processing task. Signal differences (BOLD changes) were compared between baseline and endpoint, separately for BE-SMART-DR or BE-SMART-ER, at a voxel-level threshold of p<0.001 uncorrected using statistical parametric mapping (SPM) software. If voxels above this threshold survived in a hypothesized region of interest (amygdala and ventral prefrontal cortex, VPFC) then the signal differences in those voxels were extracted and mean values within the region for each subject were used in the analyses below. The only voxel-based finding meeting criteria was left amygdala activation decreases to fearful faces in participants receiving BE-SMART-DR. The results of the mixed model analysis of those values are below.
Time Frame: baseline and 12 weeks
Population: Adolescents and young adults with bipolar disorder (BD) who received intervention and had both baseline and endpoint fMRI data of sufficient quality were analyzed. Voxel-level threshold for BE-SMART-ER did not reach p<0.001 uncorrected threshold and therefore there were no extracted values for further analyses.
Measure: Least Squares Mean (Standard Error); unit: BOLD signal
Groups:
- BE-SMART DR: Adolescents and young adults with BD who received baseline and endpoint scans and BE-SMART-DR and had fMRI activation data at both timepoints of sufficient quality for analyses.
- BE-SMART ER: Adolescents and young adults with BD who received baseline and endpoint scans and BE-SMART-ER and had fMRI activation data at both timepoints of sufficient quality for analyses.
Arm/Group | BE-SMART DR | BE-SMART ER
Number analyzed (Participants) | 11 | 0
BOLD signal
  Baseline | 1.62 (0.64) |
  12 weeks | -1.42 (0.64) |
Statistical Analysis 1: Comparison: BE-SMART DR; Test type: Other — Mixed model with time (baseline and endpoint) as within-subjects factor; compare Least Square (LS) estimate of endpoint minus baseline to zero. The best-fitting model was chosen based on information criteria; p = 0.0001, t-test, 2 sided; Endpoint minus Baseline = -3.04, 95% CI 2-sided [-4.14 to -1.93], Standard Error of Mean 0.5

2. Primary Outcome: FMRI BOLD Signal Changes in Left Amygdala at Baseline and Midpoint
Description: Signal differences (BOLD changes) between baseline and midpoint in regions of interest that survived the voxel-based threshold in participants who received either BE-SMART variation and had fMRI data of sufficient quality for fMRI activation analyses. The results of the mixed model analyses of those values are below.
Time Frame: Baseline and 6 weeks
Population: Adolescents and young adults with BD who received BE-SMART-DR and who had fMRI data at both at baseline and midpoint. Voxel-level threshold for BE-SMART-ER did not reach the p<0.001 uncorrected threshold and therefore there were no extracted values for further analyses.
Measure: Least Squares Mean (Standard Error); unit: BOLD signal
Groups:
- BE-SMART-DR: Adolescents and young adults with BD who received baseline, midpoint and endpoint scans and BE-SMART-DR and had fMRI activation data at baseline and midpoint of sufficient quality for analyses.
- BE-SMART-ER: Adolescents and young adults with BD who received Baseline, midpoint and endpoint scans and BE-SMART-ER and had fMRI activation data at baseline and midpoint of sufficient quality for analyses.
Arm/Group | BE-SMART-DR | BE-SMART-ER
Number analyzed (Participants) | 11 | 0
BOLD signal
  Baseline | 1.42 (0.75) |
  6 weeks | 0.053 (1.93) |
Statistical Analysis 1: Comparison: BE-SMART-DR; Test type: Other — Mixed model with time (baseline and midpoint) as within-subjects factor; compare LS estimate of midpoint minus baseline to zero; p = 0.60, t-test, 2 sided; Midpoint minus Baseline = -1.37, 95% CI 2-sided [-6.97 to 4.23], Standard Error of Mean 2.51

3. Primary Outcome: fMRI Functional Connectivity Changes in VPFC From an Amygdala Seed Region at Baseline and Endpoint
Description: Pearson's correlations between the mean timecourse of the seed and the timecourse of each voxel between baseline and endpoint were compared at a voxel-level threshold of p<0.001 uncorrected using statistical parametric mapping (SPM) software. If there were voxels above this threshold in the hypothesized region of interest (ventral prefrontal cortex), then the correlation values from those voxels in that region were extracted and Fisher transformed and averaged, where higher scores indicted greater connectivity. Functional connectivity differences between baseline and endpoint in regions of interest that survived the voxel-based threshold in participants who received either BE-SMART variation and had fMRI data of sufficient quality for fMRI functional connectivity analyses. The results of the mixed model analysis of those values are below.
Time Frame: Baseline and 12 weeks
Population: Only adolescents and young adults with BD who had baseline and endpoint fMRI functional connectivity data of sufficient quality were analyzed. Voxel-level threshold for BE-SMART-ER did not reach the p<0.001 uncorrected threshold and therefore there were no extracted values for further analyses.
Measure: Least Squares Mean (Standard Error); unit: Z-transformed correlation coefficient
Arm/Group | BE-SMART DR | BE-SMART ER
Number analyzed (Participants) | 11 | 0
Z-transformed correlation coefficient
  Baseline | -0.057 (0.017) |
  12 weeks | 0.052 (0.017) |
Statistical Analysis 1: Comparison: BE-SMART DR; Test type: Other — Mixed model with time (baseline and endpoint) as within-subjects factor; compare LS estimate of endpoint minus baseline to zero; p = 0.0001, t-test, 2 sided; Endpoint minus Baseline = 0.11, 95% CI 2-sided [0.074 to 0.146], Standard Error of Mean 0.016

4. Primary Outcome: fMRI Functional Connectivity Changes in VPFC From an Amygdala Seed Region at Baseline and Midpoint
Description: Pearson's correlations between the mean timecourse of the seed and the timecourse of each voxel between baseline and midpoint were compared at a voxel-level threshold of p<0.001 uncorrected using statistical parametric mapping (SPM) software. If there were voxels above this threshold in the hypothesized region of interest (ventral prefrontal cortex), then the correlation values from those voxels in that region were extracted and Fisher transformed and averaged where higher scores indicte greater connectivity. Functional connectivity differences between baseline and midpoint in regions of interest that survived the voxel-based threshold in participants who received either BE-SMART variation and had fMRI data of sufficient quality for fMRI functional connectivity analyses. The results of the mixed model analysis of those values are below.
Time Frame: Baseline and 6 weeks
Population: Adolescents and young adults with BD who received BE-SMART-DR with fMRI functional connectivity data at both baseline and midpoint. Voxel-level threshold for BE-SMART-ER did not reach the p<0.001 uncorrected threshold and therefore there were no extracted values for further analyses.
Measure: Least Squares Mean (Standard Error); unit: Z-transformed correlation coefficient
Groups:
- BE-SMART-DR: Adolescents and young adults with BD who received baseline and midpoint scans and BE-SMART-DR and had fMRI data at both timepoints of sufficient quality for functional connectivity analyses.
- BE-SMART-ER: Adolescents and young adults with BD who received baseline and midpoint scans and BE-SMART-ER and had fMRI data at both timepoints of sufficient quality for functional connectivity analyses.
Arm/Group | BE-SMART-DR | BE-SMART-ER
Number analyzed (Participants) | 9 | 0
Z-transformed correlation coefficient
  Baseline | -0.038 (0.026) |
  6 weeks | -0.0068 (0.046) |
Statistical Analysis 1: Comparison: BE-SMART-DR; Test type: Other — [test comment as in outcome 2, analysis 1]; p = 0.58, t-test, 2 sided; Midpoint minus Baseline = 0.031, 95% CI 2-sided [-0.095 to 0.157], Standard Error of Mean 0.055

ADVERSE EVENTS:
Time Frame: up to 12 weeks
Groups:
- BE-SMART: The group received Brain Emotion Circuitry-Targeted Self-Monitoring and Regulation Therapy (BE-SMART), an intervention designed to provide improvements to the functioning of emotion brain circuitry with variations that focus on either providing skills to improve explicit emotion regulation (BE- SMART-ER) or to regularize sleep and other daily rhythms (BE-SMART-DR).
  Participants took part in BE-SMART, designed to be comprised of 12 therapy sessions, at a rate of about 1 session every one to two weeks. Participants were asked to complete worksheets and practice the skills learned from the sessions and asked questions about their symptoms and behaviors. There were interview assessments and scanning performed prior to providing the intervention and at the midpoint and endpoint. The intervening 9 sessions were performed by video telecommunication. Each subject received one of two BE-SMART variations both designed to target the functioning of emotion regulation brain circuitry: one with main focus on providing skills to improve explicit emotion regulation (BE- SMART-ER) and one with main focus to regularize sleep and other daily rhythms (BE-SMART-DR).
Arm/Group | BE-SMART
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-06-15): https://cdn.clinicaltrials.gov/large-docs/88/NCT03183388/Prot_SAP_000.pdf